CLINICAL TRIAL: NCT05075889
Title: A Single-center Study Investigating the Utility of Indocyanine Green (ICG) Fluorescence Imaging in Patients With Benign Bone Tumors Requiring Intralesional Operative Management
Brief Title: Utility of ICG in Benign Bone Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Eric R. Henderson, Associate Professor of Orthopaedics, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY02000819
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Bone Tumor
Keywords: Benign; Operative Management
MeSH Terms: conditions — Bone Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: All participants will receive the same study drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Benign Bone patients (Experimental): Patients with Benign Bone tumors requiring intralesional operative management will be administered immunofluorescent indocyanine green 24 hours prior to surgery, imaging of perfused tissues will be performed at the time of tumor removal.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Enrolled subjects will receive Indocyanine Green administered the day prior to surgery during their standard-of-care preoperative appointment
  Other Names: ICG

SUMMARY:
Patients with a biopsy-proven benign bone tumor for which standard of care is intralesional operative management will receive a weight-appropriate IV dose of indocyanine green (ICG, FDA-approved) the day prior to surgery during their standard pre-operative clinic visit. On the day of surgery, fluorescence images will be obtained using a non-invasive fluorescence camera.

DETAILED DESCRIPTION:
ICG fluorescence imaging has been used to assess tissue perfusion in vivo in real-time intra-operative arterial and lymphatic perfusion imaging and osseous flap perfusion imaging. Compared to the conventional medical imaging modalities, such as computed tomography (CT) or magnetic resonance imaging (MRI), ICG fluorescence imaging is nonionizing, low-cost, and portable. ICG is a dye that absorbs near-infrared light in the wavelength range between 790 to 805 nm and has an emission at the peak of 835 nm. ICG is almost 98% plasma protein-bound so that once it is received in the microcirculation, it remains within the lymphatic and circulatory vasculature unless inflammation is present. ICG has been approved for clinical use by the Food and Drug Administration (FDA) since 1959. Since then, ICG has been used in humans for angiography in ophthalmology and cardiology applications and is given routinely to patients in these clinical settings. ICG fluorescence imaging has also been used to guide laparoscopic surgery, robotic adrenalectomy, assess tissue perfusion in vivo in real-time intra-operative arterial and lymphatic perfusion imaging, and tissue flap perfusion imaging. ICG is ideal to measure perfusion/blood flow because it binds efficiently to blood lipoproteins and thus does not leak from circulation under normal circumstances. In addition, the ICG half-life is short making repeated measures possible, and it is indirectly activated, so that the dynamic fluorescence due to bone and tissue perfusion can be captured by a video rate imaging system.

The dynamic fluorescence imaging systems to be used in this study will be preferentially the Pentero surgical microscope (Zeiss, Germany), Spy Elite Imaging System or SPY Portable Handheld Imaging (SPY-PHI) System (Novadaq/Stryker), or another imager may be used. These imagers are commercially available imaging systems that are used to assess tissue perfusion in real time in the operating room. The systems have a multi-directional imaging arm which contains a near-infrared light source that illuminates the fluorescent agent within the tissues, a high definition (HD) video camera that captures the intensity of fluorescent marker in real-time, and software that allows the user to capture relative and absolute perfusion values within the surgical field. These products are FDA-approved for use to monitor blood flow, plastic surgery, microsurgery, reconstructive surgery, gastrointestinal imaging and coronary bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 12 years of age or older
2. Diagnosis of any of the following that has been identified by imaging and/or biopsy:

   1. Enchondroma
   2. Periosteal chondroma
   3. Osteochondroma
   4. Chondroblastoma
   5. Giant cell tumor of bone
   6. Aneurysmal bone cyst
   7. Unicameral (aka Simple) bone cyst
   8. Chondromyxoid fibroma
   9. Osteoblastoma
   10. Desmoplastic fibroma
   11. Fibrous dysplasia
   12. Osteofibrous dysplasia
3. Intralesional operative management for their tumor planned
4. Written informed consent signed by the subject if 18 years of age or older or by parent(s) or legally authorized representative if younger than 18 years of age. If younger than 18 years of age, the child must be able to be assent.

Exclusion Criteria:

1. Iodine allergy
2. Women who are pregnant or breastfeeding
3. Incarcerated individuals

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Fluorescent intensity contrast | 24 hours post injection
  fluorescence contrast suitable to facilitate fluorescence-guided surgical resection of benign bone tumors (tumor-to-background ratio > 2.0)

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Henderson, MD, Principal Investigator — Dartmouth-Hithcock Medical Center
Locations (1):
- Dartmouth-Hitchock, Lebanon, New Hampshire, United States